CLINICAL TRIAL: NCT03103542
Title: A Non-Controlled, Open-Label, Multicenter, Study of Immune Tolerance Induction Performed With rFVIIIFc Within a Timeframe of 60 Weeks in Severe Haemophilia A Patients With Inhibitors Who Have Failed Previous Immune Tolerance Induction Therapies
Brief Title: Study of rFVIIIFc for Immune Tolerance Induction (ITI) in Haemophilia A Patients With Inhibitors Who Have Failed Previous ITI Therapies
Acronym: ReITIrate
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Swedish Orphan Biovitrum (Industry)
Collaborators: Bioverativ Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sobi.Elocta-003; 2017-000065-73 (EudraCT Number)
Record Dates: First submitted 2017-03-31; First posted 2017-04-06 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Hemophilia A
Keywords: ITI; rFVIIIFc; Immune Tolerance Induction
MeSH Terms: conditions — Hemophilia A | interventions — factor VIII-Fc fusion protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Recombinant coagulation factor VIII Fc (rFVIIIFc) (Experimental): Participants will receive rFVIIIFc at a dose of 200 international units (IU)/kilogram (kg) as once daily injections or divided on several injections per day at the discretion of the Investigator, starting at baseline visit up to maximum of 60 Weeks during the ITI Period. Participants who meet the criteria for ITI success will enter a tapering period of 16 weeks where the dose will be tapered down until a prophylactic dose, as judged by the Investigator, is achieved and thereafter a follow-up period of 32 weeks where the patient will continue to receive prophylactic treatment with rFVIIIFc.
  Interventions: Biological: Recombinant coagulation factor (rFVIIIFc)

INTERVENTIONS:
Biological: Recombinant coagulation factor (rFVIIIFc) — rFVIIIFc 200 IU/kg/day during ITI Period and thereafter adjusted according to the Investigator's judgement
  administered intravenously.
  Other Names: ELOCTA; ELOCTATE

SUMMARY:
The primary purpose of this study is to describe the outcome of Immune Tolerance Induction (ITI) treatment performed with rFVIIIFc within a timeframe of 60 weeks in patients with haemophilia A who have failed previous attempts at tolerization.

DETAILED DESCRIPTION:
This is an open-label, single-arm, interventional multi-center study designed to explore ITI performed with recombinant coagulation factor VIII Fc fusion protein (rFVIIIFc) within a timeframe of 60 weeks in patients with severe haemophilia A, who have failed previous attempts at tolerization including use of immunosuppressants.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent provided by the patient, or the patient's legally authorized representative for patients under the legal age. Assent should be obtained from pediatric patients according to local regulations
2. Male patients of any age diagnosed with severe haemophilia A, as confirmed from the medical record
3. Previously treated with any plasma-derived or recombinant conventional or extended half-life FVIII
4. Diagnosed with high titer inhibitors (historical peak ≥5 Bethesda units (BU)/mL according to medical records)
5. Inhibitor titer >0.6 BU at screening
6. Failed previous ITI attempt(s) with any plasma-derived or recombinant conventional or extended half-life FVIII including the use of immunosuppressant The attempt should be documented in the medical records and have the following characteristics:

   * A minimum FVIII dose equivalent to the low dose arm of the International ITI study (50 IU/kg, 3 times/week)
   * A minimum ITI treatment period of 33 months or
   * Shorter than 33 months if no downward trend of at least 20% in the inhibitor titer in a 6-month period after the initial 3 months of the ITI treatment
7. All patients must practice effective contraception during the study and for 3 months after their last dose of study treatment

Exclusion Criteria:

1. Other coagulation disorder(s) in addition to haemophilia A
2. History of hypersensitivity reactions associated with any rFVIIIFc administration
3. High risk of cardiovascular, cerebrovascular, or other thromboembolic events, as judged by the investigator
4. Planned major surgery to be deferred after study completion. Minor surgery such as tooth extraction or insertion/replacement of central venous access device is allowed.
5. Concurrent systemic treatment with immunosuppressive drugs within 12 weeks prior to screening. Exceptions to this include: ribavirin for treatment of Hepatitis C virus (HCV), and/or systemic steroids (a total of 2 courses of pulse treatments lasting no more than 7 days within 12 weeks prior to Day 1) and/or inhaled steroids
6. Abnormal renal function (serum creatinine >2.0 mg/dL) as assessed by local lab
7. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN) as assessed by local lab
8. Serum total bilirubin >3 × ULN as assessed by local lab
9. Cluster of differentiation 4 (CD4) lymphocytes ≤200 mm3 if known as HIV antibody positive at Screening
10. Viral load of ≥400 copies/mL if known HIV antibody positive at Screening
11. Patients with a documented history of alcohol or substance abuse within 12 months prior to randomization
12. Previous inclusion in this study
13. Participation in another concurrent clinical interventional study within 30 days of screening or intake of an investigational drug within five half-lives of that investigational drug has passed
14. Foreseeable inability to cooperate with given instructions or study procedures
15. Presence of any medical or psychological condition or laboratory result that in the opinion of the investigator can interfere with the patient's ability to comply with the protocol requirements or makes the patient not appropriate for inclusion to the study and treatment with rFVIIIFc

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2019-09-04 (Actual); Study Completion 2020-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Study Medical Director
Locations (12):
- Swedish Orphan Biovitrum Research Site, Washington D.C., District of Columbia, United States
- Canada (2):
  - Swedish Orphan Biovitrum Research Site, Hamilton
  - Swedish Orphan Biovitrum Research Site, Vancouver
- Germany (3):
  - Swedish Orphan Biovitrum Research Site, Bonn
  - Swedish Orphan Biovitrum Research Site, Frankfurt am Main
  - Swedish Orphan Biovitrum Research Site, Mörfelden-Walldorf
- Swedish Orphan Biovitrum Research site, Dublin, Ireland
- Swedish Orphan Biovitrum Research Site, Ljubljana, Slovenia
- Swedish Orphan Biovitrum Research site, Gothenburg, Sweden
- United Kingdom (3):
  - Swedish Orphan Biovitrum Research Site, Birmingham
  - Swedish Orphan Biovitrum Research Site, Liverpool
  - Swedish Orphan Biovitrum Research Site, London

IPD SHARING:
Plan to Share IPD: Yes
According to Sobi's data sharing policy Sobi may share anonymized clinical study data with qualified researchers. Sobi commits to sharing clinical study data on participant level and summary data for medicines and indications approved by EMA and/or FDA. Data access will be granted in response to qualified research requests. All requests are evaluated by a cross functional panel of experts within Sobi.
Time Frame: Evaluated on a case by case basis
Access Criteria: A decision on data sharing will be based on the following:
  * The scientific merit of the proposal - i.e. the proposal should be scientifically sound, ethical, and have the potential to contribute to the advancement of public health.
  * The feasibility of the research proposal - i.e. the requesting research team must be scientifically qualified and have the resources to conduct the proposed project.
  * Maintenance of personal integrity - i.e. Sobi will not consider sharing individual data if there is a risk of re-identification of individuals despite a proper anonymisation. Moreover, the patients' informed consent will always be respected. Sobi reserves the right to reject the proposal if the anonymisation process will render unusable data.
  * Publication of results - the applicants should commit to submit their findings to a peer-reviewed scientific journal, alternatively to present the results at a congress (poster or similar), regardless of the research outcome
URL: https://www.sobi.com/en/policies

REFERENCES:
- [Derived] Konigs C, Meeks SL, Nolan B, Schmidt A, Lofqvist M, Dumont J, Leickt L, Nayak S, Lethagen S. Rescue immune tolerance induction with a recombinant factor Fc-fused VIII: prospective ReITIrate study of clinical, humoral and cellular immune responses. Ther Adv Hematol. 2024 Nov 23;15:20406207241300809. doi: 10.1177/20406207241300809. eCollection 2024. PMID 39583653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was open at 18 sites in 9 countries in Northern America and Europe. 11 sites in 7 countries recruited patients. It was initially planned to enroll 20 patients but due to recruitment challenges and a changing treatment landscape the recruitment was stopped after enrolling 16 patients. Recruitment was open from Aug 2017 to Nov 2019. 18 patients were screened and 16 enrolled into this study.
Pre-assignment Details: After informed consent was provided, patients underwent study specific screening procedures. During the 4- to 6-week screening period, patients continued with their usual treatment regimen in accordance with the local standard of care. Patients who met all inclusion and no exclusion criteria specified by the protocol were enrolled into the study. The 2 screening failures did not meet inclusion criteria 1 (signed informed consent) and 5 (inhibitor titer ≥0.6 BU at screening) respectively.
Groups:
- Recombinant Coagulation Factor VIII Fc (rFVIIIFc): Participants received rFVIIIFc at a dose of 200 international units (IU)/kilogram (kg) as once daily injections or divided on several injections per day at the discretion of the Investigator, starting at baseline visit up to maximum of 60 Weeks during the ITI Period. Participants who met the criteria for ITI success entered a tapering period of 16 weeks where the dose was tapered down until a prophylactic dose, as judged by the Investigator, was achieved and thereafter a follow-up period of 32 weeks where the patient continued to receive prophylactic treatment with rFVIIIFc.
  Recombinant coagulation factor (rFVIIIFc): rFVIIIFc 200 IU/kg/day during ITI Period and thereafter adjusted according to the Investigator's judgement administered intravenously.
Period: Overall Study
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Started | 16 (18 - screened 16 - enrolled)
Completed | 9
Not Completed | 7
Not completed — Physician Decision | 2
Not completed — Adverse Event | 2
Not completed — Other | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Recombinant Coagulation Factor VIII Fc (rFVIIIFc): Participants will receive rFVIIIFc at a dose of 200 international units (IU)/kilogram (kg) as once daily injections or divided on several injections per day at the discretion of the Investigator, starting at baseline visit up to maximum of 60 Weeks during the ITI Period. Participants who meet the criteria for ITI success will enter a tapering period of 16 weeks where the dose will be tapered down until a prophylactic dose, as judged by the Investigator, is achieved and thereafter a follow-up period of 32 weeks where the patient will continue to receive prophylactic treatment with rFVIIIFc.
  Recombinant coagulation factor (rFVIIIFc): rFVIIIFc 200 IU/kg/day during ITI Period and thereafter adjusted according to the Investigator's judgement
  administered intravenously.
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants] — Age at baseline
  Participants
    <=18 years | 15
    Between 18 and 65 years | 1
    >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 7.5 [3 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 15
  Race: Asian | 0
  Race: Black or African American | 1
  Race: American Indian or Alaska Native | 0
Region of Enrollment [Number; unit: participants]
  Canada | 3
  Sweden | 1
  United States | 1
  Ireland | 3
  United Kingdom | 3
  Slovenia | 1
  Germany | 4
Hemophilia history - severity [Count of Participants; unit: Participants]
  Mild | 0
  Moderate | 0
  Severe | 16
Hemophilia history - Family history of Inhibitors [Count of Participants; unit: Participants]
  Yes | 7
  No | 5
  Unknown | 4
Number of previous ITI Treatments [Count of Participants; unit: Participants]
  1 Treatment | 10
  2 Treatments | 4
  3 Treatments | 2
Inhibitor History - Historical Peak Titre Level [Median (Full Range); unit: BU/ml] | 127.4 [8 to 3000]
Inhibitor history - Age at Inhibitor development [Mean (Standard Deviation); unit: years] | 1.9 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: ITI Success
Description: Number of patients who achieve ITI success where ITI success is defined as achieving all 3 of the following criteria:
  * Negative titer for inhibitor (<0.6 Bethesda units/mL by the Nijmegen-modified Bethesda assay) at 2 consecutive visits
  * FVIII incremental recovery (IR) >66% of the expected IR at 2 consecutive visits
  * FVIII half-life (t½) ≥7 hours
Time Frame: up to 60 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Participants
  ITI success | 1
  Partial Success | 2
  ITI failure | 6
  Not determinable due to withdrawal during the ITI | 7

2. Secondary Outcome: Time to ITI Success
Description: Time to the patient reaches ITI success according to the pre-defined criteria
  For the subset of patients who were classified as partial success at the end of the ITI period, the time to fulfillment of the criteria for partial success was also analyzed descriptively.
Time Frame: up to 60 weeks
Population: 1 patient achieved ITI success and 2 patients achieved partial success
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 3
weeks
  Time to ITI success | 46.71 (0)
  Time to Partial Success | 38.76 (15.05)

3. Secondary Outcome: Occurrence of Relapse During a 48-week Period Following Successful ITI Treatment
Description: Relapse was defined as a positive inhibitor (≥0.6 BU/mL) on 2 consecutive assessments and incremental recovery ≤66 % of the expected incremental recovery on 2 consecutive assessments
Time Frame: Up to 48 weeks
Population: Only patients achieving ITI success are included in the analysis for this endpoint. 1 patient achieved ITI success.
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Bleedings During ITI Treatment
Description: Only bleeds requiring treatment with rFVIIIFc or bypassing agents should be registered. A bleeding episode starts from the first sign of a bleed and ends no more than 72 hours after the last injection of bypassing agents or rFVIIIFc to treat the bleeding episode.
Time Frame: up to 60 weeks
Measure: Median (Full Range); unit: Annualized bleeding rate(bleedings/year)
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Annualized bleeding rate(bleedings/year) | 4.70 [0.00 to 45.66]

5. Secondary Outcome: Bleeding Rate During a 48-week Period Following Successful ITI Treatment
Description: as for outcome 4
Time Frame: up to 48 weeks
Population: Only patients achieving ITI success are included in the analysis for this endpoint. 1 patient achieved ITI success.
Measure: Median (Full Range); unit: Annualized bleeding rate(bleedings/year)
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 1
Annualized bleeding rate(bleedings/year) | 5.07 [5.07 to 5.07]

6. Secondary Outcome: Adverse Events (AEs)
Description: All observed adverse events as a measure of tolerability. (AE=adverse event, SAE=serious adverse event, TEAE=treatment emergent adverse event)
Time Frame: SAEs - approx 166 weeks AEs - approx 110 weeks
Measure: Number; unit: events
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
events
  TEAEs | 188
  Serious AEs | 21
  Serious TEAEs | 18
  Non-serious TEAEs | 170
  Related TEAEs | 2
  Mild AEs | 145
  Moderate AEs | 42
  Severe AEs | 4
  AEs Leading to Withdrawal | 3
  AEs Leading to Death | 0

7. Secondary Outcome: Consumption of rFVIIIFc
Description: Consumption will be assessed based on amount of administered study treatment during the ITI period.
Time Frame: Up to 60 weeks
Measure: Median (Full Range); unit: IU
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
IU | 1902625.0 [605000.0 to 7555750.0]

8. Secondary Outcome: Consumption of rFVIIIFc
Description: Consumption will be assessed based on amount of administered study treatment during the ITI period.
Time Frame: Up to 60 weeks
Measure: Median (Full Range); unit: IU/kg
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
IU/kg | 62586.7 [24226.7 to 89724.2]

9. Secondary Outcome: Number of Days Missed School or Work During ITI Treatment
Description: Days missed school or work will be registered by the patients in an electronic diary
Time Frame: up to 60 weeks
Measure: Median (Full Range); unit: Days/year
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Days/year | 0.5 [0 to 59]

10. Secondary Outcome: Number of Days Missed School or Work During ITI Treatment
Description: Days missed school or work will be registered by the patients in an electronic diary
Time Frame: up to 60 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Days | 0.5 [0 to 50]

11. Secondary Outcome: Number of Days Missed School or Work During a 48-week Period Following Successful ITI Treatment
Description: Days missed school or work will be registered by the patients in an electronic diary
Time Frame: up to 48 weeks
Population: Only patients achieving ITI success are included in the analysis for this endpoint. 1 patient achieved ITI success.
Measure: Median (Full Range); unit: Days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 1
Days | 0 [0 to 0]

12. Secondary Outcome: Number of Hospitalizations During ITI Treatment
Description: Days of hospitalization will be collected by the Investigator at the study visits
Time Frame: up to 60 weeks
Measure: Median (Full Range); unit: Days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
Days | 0 [0 to 36]

13. Secondary Outcome: Number of Hospitalizations During a 48-week Period Following Successful ITI Treatment
Description: Days of hospitalization will be collected by the Investigator at the study visits
Time Frame: Up to 48 weeks
Population: Only patients achieving ITI success are included in the analysis for this endpoint. 1 patient achieved ITI success.
Measure: Number; unit: Days
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 1
Days | 0

14. Secondary Outcome: Adherence
Description: Defined as percentage of administered doses versus planned doses
Time Frame: up to 108 weeks
Population: 16 patients analyzed for the ITI period. 1 patient analyzed for the tapering and follow-up period (1 patient achieved ITI success and entered tapering and follow-up periods).
Measure: Mean (Standard Deviation); unit: % of administered vs planned doses
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
Number analyzed (Participants) | 16
% of administered vs planned doses
  ITI period | 92.52 (13.86)
  Tapering period | 100.5 (0)
  Follow-up period | 98.56 (0)

ADVERSE EVENTS:
Time Frame: SAEs: From signature of the informed consent form to the safety follow-up visit (approximately 116 weeks). Non-serious AEs: From the time of first dose of IMP to the safety follow-up visit (approximately 110 weeks).
Description: The investigator were to report all directly observed adverse events, and all adverse events spontaneously reported by the patient. In addition, each patient were to be questioned about AEs at each study visit.
  AEs are reported on overall level. Please note the difference in the reporting period of SAEs and non-serious AEs (SAEs also collected during screening period). 18 patients entered screening, 16 patients were eventually enrolled and are included in the analysis.
Arm/Group | Recombinant Coagulation Factor VIII Fc (rFVIIIFc)
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc (rFVIIIFc) (N=16)
Brachiocephalic vein thrombosis (Vascular disorders) | 1 (1)
Vena cava thrombosis (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tonsillitis (Infections and infestations) | 2 (2)
Vascular device infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (5)
Device related sepsis (Infections and infestations) | 1 (1)
Staphylococcal infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Coagulation Factor VIII Fc (rFVIIIFc) (N=16)
Haemorrhage (Vascular disorders) | 1 (1)
Seasonal allergy (Immune system disorders) | 1 (1)
Catheter site irritation (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (2)
Influenza like illness (General disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (4)
Pyrexia (General disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Autism spectrum disorder (Psychiatric disorders) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (15)
Fall (Injury, poisoning and procedural complications) | 3 (4)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (2)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 (1)
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood urine present (Investigations) | 2 (2)
Haematocrit decreased (Investigations) | 1 (1)
Haemoglobin decreased (Investigations) | 1 (1)
Human rhinovirus test positive (Investigations) | 1 (1)
Protein urine present (Investigations) | 1 (2)
Red blood cell count decreased (Investigations) | 1 (1)
Tri-iodothyronine free increased (Investigations) | 1 (1)
Urine ketone body present (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Investigations) | 1 (2)
Rhinorrhoea (Investigations) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 1 (2)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (7)
Jugular vein occlusion (Nervous system disorders) | 1 (1)
Migraine (Nervous system disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Anal incontinence (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Lip ulceration (Gastrointestinal disorders) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Tooth development disorder (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (3)
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis in device (Product Issues) | 1 (1)
Device damage (Product Issues) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (9)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Growing pains (Musculoskeletal and connective tissue disorders) | 1 (1)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1 (1)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Impetigo (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 5 (10)
Rhinitis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 3 (5)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-02-26): https://cdn.clinicaltrials.gov/large-docs/42/NCT03103542/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT03103542/SAP_001.pdf